CLINICAL TRIAL: NCT05094583
Title: The SmokeFree App Smoking Cessation Study
Acronym: SMOKEFREE
Status: Suspended | Type: Observational
Why Stopped: Suspended due to COVID19 pandemic.
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W19/044
Record Dates: First submitted 2021-02-09; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Smoking Cessation; Smoking; Smoking Reduction; Smoking Habit
Keywords: Acute Assessment Unit; Ambulatory Emergency Care
MeSH Terms: conditions — Smoking Cessation; Smoking; Smoking Reduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Arm: Patients who expressed wish to quit smoking and accept use of the SmokeFree app
  Interventions: Behavioral: Use of SmokeFree app
- Control Arm: Patients who expressed wish to quit smoking but declines all support or use of SmokeFree app

INTERVENTIONS:
Behavioral: Use of SmokeFree app — Intervention Arm
  Groups: Intervention Arm

SUMMARY:
SmokeFree is a theory-driven and evidence-based stop smoking mobile application. Based on NICE guidance and best practice for smoking cessation, the application employs over 30 behaviour change techniques used in NHS Stop Smoking Services. It has been downloaded over 4 million times and has an average user rating of 4.7 out of 5, from over 120,000 ratings. Whilst user feedback has been highly positive, there is a need for further objective studies to demonstrate its efficacy.

This is a prospective, observational, two arm feasibility study, which aims to evaluate the efficacy, attrition rate and user experience of the SmokeFree App.

Inpatients in the Acute Medical Unit and ambulatory emergency care unit at Chelsea and Westminster Hospital who are current smokers will be offered to participate in the study, in addition to all other smoking cessation interventions, which will also be offered to them. Care will be taken to ensure that all available options of smoking cessation support are offered in addition to the SmokeFree application. Subjects agreeing to participate will be given access to the application for a period of 12 weeks, with a target quit date no later than week 8 of use of the application. At the end of 12 weeks they will be offered a follow up appointment in a purposely designed clinic, where their CO level will be measured, as well as being invited to complete feedback questionnaires on their experience.

The primary end point of the study will be the quit rate for a period of minimum of 4 weeks by the completion of the 12 week trial. This will be confirmed with exhaled carbon monoxide testing.

Secondary endpoints include user experience, engagement with the mobile application and attrition rate.

ELIGIBILITY:
Inclusion Criteria:

Intervention:

* ≥ 18 years
* All new patients admitted via the Acute medical via AAU (or AEC)
* Current smoker and willing to quit
* Smartphone owner
* Fluent in English (verbal and written)
* Able to give informed consent
* Able and willing to attend a follow up visit in 12 weeks.

Control:

- Meet above inclusion criteria except ownership of smartphone.

Exclusion Criteria:

* < 18 years
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participant will be recruited from the Acute Assessment Unit and Ambulatory Emergency Care at Chelsea and Westminster Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-12-04 (Estimated); Study Completion 2021-12-04 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence | 12 weeks
  Percentage of participants who achieved sustained abstinence over 4 weeks, within 12 weeks from starting to use the SmokeFree app, compared against outcomes for patients who expressed wish to quit but declined use of the SmokeFree app (This will be confirmed with CO testing at 12-week follow-up visit).

OTHER OUTCOMES:
User experience | 12 weeks
  User experience - measured with usability survey completed by intervention arm subjects at 12-week follow-up visit.
Attrition rate | 12 weeks
  Percentage of patients enrolled in the intervention arm, who complete the full 12 weeks of treatment
Level of engagement with the SmokeFree app | 12 weeks
  Number of log in sessions and average time spent using the SmokeFree app per session

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, Lonson, United Kingdom

DOCUMENTS (1):
  • Informed Consent Form (2019-09-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT05094583/ICF_000.pdf